CLINICAL TRIAL: NCT02231203
Title: Effect of Intravenous Omega-3 Fatty Acids on the Perioperative Immune Response and Erythrocyte Function in Patients With Colon Cancer
Brief Title: Effect of Omega-3 Fatty Acids on the Perioperative Immune Response and Erythrocyte Function
Acronym: EMPIRE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical Center Alkmaar (Other)
Responsible Party: Principal Investigator, Alexander P.J. Houdijk, Dr., Medical Center Alkmaar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NL46230.029.13
Record Dates: First submitted 2014-07-29; First posted 2014-09-04 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Colon Cancer
Keywords: fish oil; omega-3 fatty acids; postoperative inflammatory response; erythrocyte function
MeSH Terms: conditions — Colonic Neoplasms | interventions — fish oil triglycerides; Fatty Acids, Omega-3; Antioxidants

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 2 infusions of NaCl, 2 ml/kg, one the night before operation and one the day after operation.
  Interventions: Drug: Placebo
- Omegaven (Active Comparator): 2 infusions of 2ml/kg, one the night before surgery and one the day after surgery
  Interventions: Drug: Omegaven

INTERVENTIONS:
Drug: Omegaven — 2 infusions, 2 ml/kg, one the night before operation and one the day after operation
  Other Names: purified fish oil; omega-3 fatty acids; eicosapentaenoicacid (EPA); docosahexaenoicacid (DHA); dl-a- tocopherol (antioxidant); Omegaven-Fresenius
  Arms: Omegaven
Drug: Placebo — 2 infusions, 2 ml/kg, one the night before operation and one the day after operation
  Other Names: NaCl 0,9%; Natriumchloride 0,9%; glass container NaCl 0,9% Fresenius Kabi
  Arms: Placebo

SUMMARY:
Ideally, the postoperative inflammatory response is part of a well-orchestrated mechanism that contributes to tissue healing and rapid recovery. An exaggerated uncontrolled inflammatory response, however may lead to catabolism, tissue damage and organ failure. Omega-3 fatty acids may provide a means to alter cellular immune responses to the benefit of the patient. When omega-3 fatty acids are incorporated into membranes of inflammatory cells, they trigger intracellular signalling pathways that result in a less pro-inflammatory response. They modify gene and protein expression, modulate membrane protein activity and act as a reservoir for bioactive molecules. They also have a strong anti-inflammatory effect by mediating resolution of the inflammation. Furthermore, omega-3 fatty acids improve erythrocyte function, which is vital for an adequate microcirculation, tissue oxygenation and wound healing.

The investigators hypothesize that the perioperative administration of intravenous omega-3 fatty acids results in a rapid incorporation in immune cells and erythrocytes, thereby reducing the postoperative inflammatory response and improving erythrocyte function in patients undergoing colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male or female) undergoing elective laparoscopic surgery for colon cancer
* Age between 60 and 80 years
* BMI between 20 kg/m2 and below 30 kg/m2
* Written informed consent

Exclusion Criteria:

* Participation in or having participated in another clinical trial within the previous 3 months
* Indications for continuously use of anticoagulant medication and no possibility to stop these medication perioperatively, for example patients with an artificial heart valve
* Pre-operative Hemoglobin<5.0 mmol/L
* Metastatic disease
* Very poor peripheral venous access
* Current history of inflammatory or infectious disease
* The use of anti-inflammatory drugs
* The use of thyroid medication
* The use of fish oil products or fish consumption more than 2 times a week
* Contra-indication for the use of Omegaven-Fresenius, including:
* General contra-indications for parenteral nutrition
* Allergy to fish or egg protein.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in ex vivo production of pro-inflammatory cytokine IL-6 in LPS stimulated whole blood | baseline, day of surgery, postoperative day 1,2 and 4
  Ex vivo stimulation of whole blood with LPS (lipopolysaccharide, component of gram negative bacteria) resulting in the production of the pro-inflammatory cytokine IL-6, measured in ng/ml.

SECONDARY OUTCOMES:
Change in ex vivo production of TNF-α and IL-10 in LPS stimulated whole blood | baseline, day of surgery, postoperative day 1, 2 and 4
  Ex vivo stimulation of whole blood with LPS (lipopolysaccharide, component of gram negative bacteria) resulting in the production of the pro-inflammatory cytokine TNF-α (tumor necrosis factor-α), and the anti-inflammatory cytokine IL-10 (interleukine-10), both measured in ng/ml.
Change in erythrocyte function | baseline, day of surgery, postoperative day 1, 2 and 4
  Erythrocyte deformability and aggregation measured by LORRCA (laser assisted optical rotational red cell analyzer)
Change in in vivo systemic inflammatory response parameters | baseline, day of surgery, postoperative day 1, 2 and 4
  White blood cell count, C-reactive protein and cytokine levels (Interleukine-6, Tumor Necrosis Factor-α and Interleukine-10) in serum.

OTHER OUTCOMES:
Postoperative outcome (composite measure of length of stay and complications) | Registration during admission, follow up 2 and 4 weeks after surgery
  Length of hospital stay and occurence of surgical site infection, abscess, urinary tract infection, pneumonia, anastomotic leakage, need for Intensive Care Unit admission, Systemic Inflammatory Response Syndrome, Multi Organ Failure, any adverse events.
Cognitive function | baseline, follow up 2 weeks after surgery
  Neuropsychological examination using a reading test, an auditory verbal learning test, WAIS III figure series and trail making tests.

CONTACTS AND LOCATIONS:
Overall Officials: A.P.J. Houdijk, Dr., Principal Investigator — Medical Center of Alkmaar
Locations (1):
- Medical Center of Alkmaar, Alkmaar, North Holland, Netherlands

REFERENCES:
- [Derived] Bakker N, van den Helder RS, Stoutjesdijk E, van Pelt J, Houdijk APJ. Effects of perioperative intravenous omega-3 fatty acids in colon cancer patients: a randomized, double-blind, placebo-controlled clinical trial. Am J Clin Nutr. 2020 Feb 1;111(2):385-395. doi: 10.1093/ajcn/nqz281. PMID 31826232